CLINICAL TRIAL: NCT00225446
Title: Computer-Assisted Orthognathic Surgery With a Third Generation Optic Repositioning System.
Brief Title: Micron Tracker: Computer-Assisted Orthognathic Surgery With a Third Generation Optic Repositioning System
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Eric Svahn, University Hospital Grenoble
Allocation: Non-Randomized | Model: Single Group | Masking: Double
Other Study IDs: DCIC 04 14
Record Dates: First submitted 2005-09-22; First posted 2005-09-23 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Computer-Assisted Surgery; Maxillofacial Surgery
Keywords: Orthognathic surgery.; optic repositioning system.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Device: MicronTracker — MicronTracker is a Third Generation Optic Repositioning System in orthognatic surgery.

SUMMARY:
The main objective of this study is to validate a simplified platform of a repositioning system in orthognathic surgery (a third generation optic repositioning system called MicronTracker) compared with the actual clinically validated one (Orthopilot system).

DETAILED DESCRIPTION:
For the past 10 years, the use of computer-assisted surgery has expanded and is now widely spread in the orthopaedic domain, but not in maxillary-facial surgery. The main disadvantages of this technique are the necessity to fix a mark on the eyebrow with two transcutaneous pins, which is a long and invasive act, and to connect the infrared transmitter which is in contact with the patient with the computer in a limited surgery area. In this study, we want to show that the new repositioning optic systems are performing similarly to the actual validated one, that they permit to suppress the transcutaneous pins and the computer connection, and that it reduces the financial cost of this surgery. Neither the surgery technique, nor the pre-operative check-up will be modified in the study. The two repositioning systems will be used simultaneously during the mandibular osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular orthognathic surgery

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
spatial coordinates of the target (3 translations and 3 rotations) | during surgery

SECONDARY OUTCOMES:
time to install the eyebrow mark with each technique. | during surgery
adverse events due to the transcutaneous pins. | during surgery
number of handling realized by the nurse for each technique. | during surgery
evaluation of cost: number of cable versus number of marker. | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Georges BETTEGA, M.D., Ph.D., Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Maxillofacial and Plastic Surgery Department - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Bettega G, Cinquin P, Lebeau J, Raphael B. Computer-assisted orthognathic surgery: clinical evaluation of a mandibular condyle repositioning system. J Oral Maxillofac Surg. 2002 Jan;60(1):27-34; discussion 34-5. doi: 10.1053/joms.2002.29069. PMID 11757002
- [Background] Bettega G, Dessenne V, Raphael B, Cinquin P. Computer-assisted mandibular condyle positioning in orthognathic surgery. J Oral Maxillofac Surg. 1996 May;54(5):553-8. doi: 10.1016/s0278-2391(96)90630-8. PMID 8632238
- [Background] Dessenne V. Gestes médico-chirurgicaux assistés par ordinateur: applications à la ligamentoplastie du genou et à la chirurgie orthognatique. Thèse de Génie biologique et médical, Grenoble 1996
- [Background] Bettega G. La chirurgie orthognatique assistée par ordinateur: de la planification à la réalisation. Thèse de Génie biologique et médical, Grenoble 1997